CLINICAL TRIAL: NCT06215027
Title: Os Efeitos da dança Como Recurso terapêutico em Pacientes Com câncer de Mama Submetidas a Tratamento cirúrgico
Brief Title: The Effects of Dance for Breast Cancer Patients Undergoing Surgical Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Leticia Zumpano Cardenas, PHD, physiotherapist at the intensive care unit, stricto sensu postgraduate professor, AC Camargo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 74502023.7.0000.5432
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance (Experimental): Dance
  Interventions: Other: Dance

INTERVENTIONS:
Other: Dance — Dance protocol

SUMMARY:
The goal of this non randomized clinical trial, with pre- and post-intervention evaluation, longitudinal, with prospective data collection is to evaluate the effects of dance as a therapeutic intervention in breast cancer patients undergoing surgical treatment.

DETAILED DESCRIPTION:
The hypothesis is that dance will promote improvements in range of motion, strength, fatigue, functionality, pain and quality of life for breast cancer patients undergoing surgical treatment. Objectives: To evaluate the effects of dance as a therapeutic intervention in breast cancer patients undergoing surgical treatment on: shoulder range of, overall muscle strength, fatigue, respiratory muscle strength, functionality, pain and quality of life. Method: This is a non-randomized randomized clinical trial, with pre- and post-intervention evaluation, prospective data collection. The following will be used for pre-intervention assessment: goniometry, dynamometry, manovacuometry, 6-minute walk test, fatigue and quality of life questionnaire, and quality of life questionnaire, as well as a pain assessment scale. After 16 weeks, the same variables will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with breast cancer
* undergone surgical resection
* after medical referral for physiotherapy
* and physiotherapeutic assessment

Exclusion Criteria:

* patients with another previous oncological diagnosis
* previous neuromuscular diseases
* patients who do not agree to take part in the study
* or the impossibility of carrying out the muscle strength assessment and/or other assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
ROM | Pre-intervention and after 16 weeks
  Shoulder range of motion

SECONDARY OUTCOMES:
Overall muscle strength | Pre-intervention and after 16 weeks
  Dynamometer
Fatigue | Pre-intervention and after 16 weeks
  Brief Fatigue Inventory. The BFI is a scale with 11 points (0 to 10), including a dichotomous question about whether the patient felt tired or fatigued in the last 7 days. For each question, zero is considered ''no fatigue'' and 10 is ''worst fatigue possible,'' except for the dichotomous question that is not scored. Among the other questions, 3 measures the severity of fatigue in the current, daily situations, and in the last 24 hours. Six questions measure the influence of fatigue in general activities, mood, walk, work, relationship with other people, and recreation. The total score is the average of all questions. According to the total score, fatigue is classified as mild (1 to 3 points), moderate (4 to 6 points), and severe (7 to 10 points).
respiratory muscle strength | Pre-intervention and after 16 weeks
  Maximum inspiratory and expiratory pressures (MIP and MEP)
Functionality | Pre-intervention and after 16 weeks
  6 minute walk test (6MWT)
Pain intensity | Pre-intervention and after 16 weeks
  Analogic visual scale. The visual analogue pain scale is a measure of pain intensity that has been widely used in several languages. For pain intensity, the scale is most commonly ranging from "no pain" (score of 0) to "worst pain imaginable" (score of 10). A higher rating indicates greater pain intensity.
Quality of life (physical well-being, social and family well-being, emotional well-being, functional well-being) | Pre-intervention and after 16 weeks
  Functional Assessment of Cancer Therapy-Breast (FACT-B). The FACT-B, version 4, is a multidimensional questionnaire composed of 37 questions divided into five domains that assess different dimensions: physical well-being, social and family well-being, emotional well-being, functional well-being and breast cancer subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Letícia Cardenas, PHD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT06215027/Prot_000.pdf